CLINICAL TRIAL: NCT05468021
Title: Puerto Rico COVID-19 Vaccine Uptake Study
Acronym: PR-COVACUPS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Puerto Rico (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Vivian Colon, Professor at the University of Puerto Rico and Researcher at the Comprehensive Cancer Center., University of Puerto Rico
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 3U54MD007600 (NIH); 3U54MD007600 (NIH)
Record Dates: First submitted 2022-07-08; First posted 2022-07-21 (Actual); Last update posted 2022-12-16 (Actual); Status verified 2022-12

CONDITIONS: COVID-19
Keywords: COVID-19 booster vaccine hesitancy; Educational intervention; COVID-19
MeSH Terms: conditions — COVID-19 | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: Participants are assigned to one of two groups in parallel for the duration of the study. 193 participants will be assigned to an educational intervention group and 193 will be assigned to a control group.
Who Masked: Participant
Masking Description: The participants will not be aware if they are assigned to an educational intervention nor control group. All will be assessed equally.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Comparison control (No Intervention): The control condition will consist of standard of care. The participants in the control arm will not receive the educational intervention after assessment.
- Intervention condition (Experimental): The participants in the intervention arm will receive the educational intervention after assessment.
  Interventions: Other: Educational intervention

INTERVENTIONS:
Other: Educational intervention — Randomized Clinical Trial (study design) to evaluate the effectiveness of an educational intervention to increase vaccine uptake among socioeconomically disadvantaged adults. The intervention will consist of a health promoter with an educational toolkit addressing misinformation, distrust, and hesitancy regarding the COVID-19 vaccine. An educational website with videos addressing COVID-19 vaccine will be available to study participants to boost information provided in the educational toolkit.
  Arms: Intervention condition

SUMMARY:
The purpose of this study is to recruit a total of 386 participants to evaluate the effectiveness of an educational program to increase the proportion of men and women aged 21 years and older who have received the COVID-19 booster vaccine

DETAILED DESCRIPTION:
This study will address vaccine hesitancy, evaluating the intervention's efficacy in a group of vulnerable and economically disadvantaged population in PR. Randomized Clinical Trial (study design) to evaluate the effectiveness of an educational intervention to increase vaccine uptake among socioeconomically disadvantaged adults. A total sample of 386 participants will be recruited. The duration of the study will consist of 1.5 hours for intervention group and 1 hour for control group.

Eligibility criteria for the study include the following: (1) age 21 years and older, (2) resident of Puerto Rico, (3) to be fully vaccinated (received the one-dose Jansen/Johnson & Johnson vaccine, -OR- received both doses of the two-dose Pfizer or Moderna vaccine), have not received booster doses against COVID-19, (4) no history of allergic reactions to any vaccine, (5) no history of mental health conditions that impede participation in the study, and (6) able to read, write, and understand Spanish.

ELIGIBILITY:
Inclusion Criteria:

1. age 21 years and older
2. resident of Puerto Rico
3. to be fully vaccinated (received the one-dose Jansen/Johnson & Johnson vaccine, -OR- received both doses of the two-dose Pfizer or Moderna vaccine)
4. have not received booster doses against COVID-19
5. no history of allergic reactions to any vaccine,
6. no history of mental health conditions that impede participation in the study
7. able to read, write, and understand Spanish.

Exclusion Criteria:

1. age 20 years and younger
2. not a resident of Puerto Rico
3. not to be fully vaccinated (have not received the one-dose Jansen/Johnson & Johnson vaccine, -OR- have not received both doses of the two-dose Pfizer or Moderna vaccine)
4. have received booster doses against COVID-19
5. history of allergic reactions to any vaccine,
6. history of mental health conditions that impede participation in the study
7. not be able to read, write, and understand Spanish.

Ages: 21 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 394 (Actual)
Dates: Start 2022-06-26 (Actual); Primary Completion 2023-06 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Rate of COVID-19 vaccine completion | Up to 4 months
  The investigators will record the vaccine brand of primary (Pfizer, Moderna, or Johnson & Johnson) and capture the vaccine administration's completion (if necessary).
Rate of COVID-10 booster vaccine uptake | Up to 4 months
  The investigators will capture the booster vaccine administration and record the vaccine brand (Pfizer, Moderna, or Johnson & Johnson).

SECONDARY OUTCOMES:
Participant's willingness to get vaccinated against COVID-19 | Up to 4 months
  Willingness to vaccinate against COVID-19 (vaccine confidence, vaccine convenience, vaccine complacency, and vaccine attitudes and beliefs), and receive the physician's recommendation to be vaccinated
Educational tool utilization by the participants | Up to 4 months
  Evaluate if participant read the educational tool

CONTACTS AND LOCATIONS:
Overall Officials: Emma Fernandez-Repollet, Ph D, Principal Investigator — Deanship of Academic Affairs RCMI Center for Collaborative Research in Health Disparities
Locations (2):
- Puerto Rico (2):
  - Outpatient Clinic, School of Medicine, University of Puerto Rico, San Juan
  - University District Hospital, San Juan